CLINICAL TRIAL: NCT07376291
Title: Use of Anti-CD146 Autoantibodies for the Diagnosis of Pulmonary Diseases Secondary to Occupational Exposure to Silica
Acronym: CD146-SILICE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-A02509-38
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Exposure Occupational; Pulmonary Diseases
Keywords: silica; Exposure occupational; Pulmonary diseases
MeSH Terms: conditions — Lung Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-exposed (Other): Subject with low exposure to silica <0.1 mg/m3 in the course of their professional activity
  Interventions: Other: Respiratory function testing; Biological: blood sampling
- Exposed (Other): Subject with moderate or high exposure to silica (>= 0.1 mg/m3) in the course of their professional activity
  Interventions: Other: Respiratory function testing; Biological: blood sampling; Radiation: CT scan

INTERVENTIONS:
Other: Respiratory function testing — Spirometry, plethysmography, FeNO test
Biological: blood sampling — 25mL peripheral blood will be collected
Radiation: CT scan — Non-injected thoracic CT scan
  Arms: Exposed

SUMMARY:
This prospective, multicenter study aims to evaluate the relevance of anti-CD146 autoantibodies (AACD146) as biological markers for the early diagnosis of pulmonary diseases related to occupational exposure to silica. Silica exposure is a recognized risk factor for fibrotic, inflammatory, and cancerous respiratory diseases. Currently, no specific biological marker exists. The hypothesis is that AACD146 reflects early effects of silica exposure. The study will include 110 participants divided into two groups (exposed vs. non-exposed) and will compare AACD146 prevalence according to exposure level and the presence of respiratory diseases.

ELIGIBILITY:
Inclusion Criteria for non-exposed group:

* Subject, male or female, aged 18 or over
* Subject with low exposure to silica <0.1 mg/m3 in the course of their professional activity, quantified during an occupational health consultation using an employment-exposure matrix
* Subjects capable of consenting to participate in the study by signing a written informed consent form
* Subjects who are beneficiaries of or affiliated with a social security system

Inclusion Criteria for exposed group:

* Subject, male or female, aged 18 or over
* Subject with moderate or high exposure to silica (>= 0.1 mg/m3) in the course of their professional activity, quantified during an occupational health consultation using an employment-exposure matrix.
* Subjects capable of consenting to participate in the study by signing a written informed consent form
* Subjects who are beneficiaries of or affiliated with a social security system

Exclusion Criteria for each group:

* Minor subject
* Subject refusing to undergo the examinations required by the protocol
* Contraindications to respiratory function tests: Recent eye or throat surgery, recent myocardial infarction or pulmonary embolism, poorly controlled high blood pressure, recent pneumothorax.
* Pregnant or breastfeeding women, patients under guardianship or curatorship, deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence ratio of AACD146 between the exposed and non-exposed groups. | At enrollment

SECONDARY OUTCOMES:
AACD146 prevalence in patients with interstitial or neoplastic lung disease. | At enrollment
AACD146 Prevalence by type of interstitial lung disease | At enrollment
AACD146 Prevalence by type of histological type of lung cancer. | At enrollment
Correlation between AACD146 and exposure duration and dose to silica | At enrollment
Correlation between AACD146 and soluble CD146 | At enrollment